CLINICAL TRIAL: NCT03855761
Title: Improving Equitable Care With Narrative Medicine and a Novel Community-based Occupational Therapy Care Model
Brief Title: Testing a Novel Community-based Occupational Therapy Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Eskenazi Health (Other)
Responsible Party: Principal Investigator, Sally Wasmuth, Principal Investigator, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: swasmuth
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Mental Disorders, Severe
MeSH Terms: conditions — Mental Disorders | interventions — Occupational Therapy; Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Experimental Occupational Therapy services
  Interventions: Behavioral: Occupational Therapy
- Comparison group (Active Comparator): Treatment as usual
  Interventions: Behavioral: Case management; psychological services

INTERVENTIONS:
Behavioral: Occupational Therapy — Detailed narrative assessment and person-centered participation in meaningful activities
  Arms: Intervention group
Behavioral: Case management; psychological services — Weekly consultation with case managers to address housing and therapy needs
  Arms: Comparison group

SUMMARY:
This study will perform a needs assessment within an outpatient mental health unit, deliver an occupational therapy model of care, track patient and organizational outcomes, and provide training to staff to implement the model.

DETAILED DESCRIPTION:
In this project the investigators' overall objective is to implement a narrative medicine-based occupational therapy (OT) model of care that brings client voices to the forefront of treatment planning and intervention to enhance the existing interdisciplinary system of service delivery within Midtown Community Mental Health (MCMH). The investigators hope to accomplish this objective via the following specific aims:1) Assess current programming - particularly processes surrounding client assessment, treatment planning, intervention, care-coordination/residential placement, and discharge - within MCMH sites to better understand limitations/gaps previously identified by the site manager that impact equitable and effective treatment 2) Adapt an existing care model - the Art of Healing Wellness Model (AoHW) - to meet the needs of MCMH, implement the model using an OT practitioner, and track feasibility/acceptability outcomes. 3) Re-assess MCMH programming post implementation to identify/demonstrate change resulting from the model 4) Using OT in the role of consultant, offer training to current MCMH staff to enable implementation of the adapted AoHW by MCMH (baccalaureate level) care coordinators 5) Preliminarily evaluate usability of the adapted AoHW by MCMH staff via focus groups following training and staff implementation

ELIGIBILITY:
Inclusion Criteria

• Patient on a pre-determined treatment team at the outpatient mental health recruitment site

Exclusion Criteria

* Under 18
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Occupational Circumstances Assessment Interview & Rating Scale (OCAIRS) | 12 weeks
  The "Occupational Circumstances Assessment Interview and Rating Scale" is a semi-structured interview that measures a person's current participation in life in 12 areas:roles, habits, personal causation, values, interests, skills, short-term goals, long-term goals, interpretation of past experiences, physical environment, social environment, & readiness for change. The assessment provides an overall quantitative summed score of participation ranging from 12 to 48 with a higher number indicating greater participation as well as individual scores of 1-4 for each subsection.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskenazi - Midtown Community Mental Health (James Wright Center), Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No